CLINICAL TRIAL: NCT07003321
Title: Study on Efficacy and Safety of HRS-4508 in Subjects With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: A Trial of HRS-4508 in Subjects With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-4508-201
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-4508 tablet (Experimental)
  Interventions: Drug: HRS-4508 tablet

INTERVENTIONS:
Drug: HRS-4508 tablet — HRS-4508 tablet

SUMMARY:
The study is being conducted to evaluate the efficacy, safety, and ORR of HRS-4508 in subjects with locally advanced or metastatic non-small cell lung cancer; Evaluate the pharmacokinetic (PK) characteristics of HRS-4508 and other efficacy endpoints for the treatment of locally advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 80 years old; Both men and women are welcome;
2. Locally advanced or metastatic non-small cell lung cancer that has failed standard treatment or cannot tolerate standard treatment regimens.
3. ECOG ratings of 0 or 1.
4. Expected survival period ≥ 12 weeks.
5. At least one measurable lesion outside the central nervous system that meets the RECIST v1.1 standard definition.
6. Willing to participate and comply with the requirements of the research protocol, and willing to cooperate with follow-up visits.

Exclusion Criteria:

1. Accompanied by untreated or active central nervous system (CNS) tumor metastasis. Subjects with a history of meningeal metastasis or current meningeal metastasis
2. There have been significant severe infections and major surgeries in the past 4 weeks
3. Existence of previous or concurrent malignant tumors
4. Difficult to treat nausea, vomiting, or other gastrointestinal diseases that affect the use of oral medication
5. Having undergone major surgeries other than diagnosis or biopsy within 28 days prior to the first administration; Experiencing traumatic minor surgery within 7 days prior to the first administration of medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events (AE)/serious adverse events (SAE) (rated based on CTCAE v5.0) | 2 years
Objective response rate (ORR) | 1 year

SECONDARY OUTCOMES:
Blood concentrations of HRS-4508 | 12 weeks
Duration of response (DoR) | 1 year
Disease control rate (DCR) | 1 year
Progression free survival (PFS) | 1 year
Overall survival (OS) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided